CLINICAL TRIAL: NCT02619188
Title: Pregnancy Unique Questionnaire of Emesis (PUQE) Methode Evaluation; Relation Between Rate of Nausea/Vomiting in Pregnancy (PUQE-score), Self-reported Nutritional Intake and Biochemical Nutritional Markers
Brief Title: Nutritional Markers in Normal and Hyperemesis Pregnancies
Acronym: PUQE-M
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Haukeland University Hospital (Other)
Collaborators: University of Bergen (Other)
Responsible Party: Sponsor
Other Study IDs: 2015/894
Record Dates: First submitted 2015-09-09; First posted 2015-12-02 (Estimated); Last update posted 2016-10-05 (Estimated); Status verified 2016-10

CONDITIONS: Hyperemesis Gravidarum; Pregnancy
Keywords: Nutrition; Hyperemesis gravidarum; Prealbumin; Questionnaire
MeSH Terms: conditions — Hyperemesis Gravidarum

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Hyperemesis gravidarum: Hyperemesis gravidarum patients admitted to hospital PUQE-form inclusion (PUQE-score), Nutritional form inclusion, Blood sampling inclusion (Prealbumin analysis), Intervention at discharge : PUQE-form, Nutritional form and Blood sampling
  Interventions: Other: PUQE-form inclusion; Other: Nutritional form inclusion; Other: Blood sampling inclusion; Other: Intervention at discharge
- Control: Healthy pregnant women: Outpatients NOT subjected to severe nausea and emesis (PUQE-score <13). PUQE-form inclusion (PUQE-score), Nutritional form inclusion, Blood sampling inclusion (Prealbumin analysis).
  Interventions: Other: PUQE-form inclusion; Other: Nutritional form inclusion; Other: Blood sampling inclusion

INTERVENTIONS:
Other: PUQE-form inclusion — PUQE-form encompassing last 24 hours completion
  Other Names: Pregnancy Unique Questionnare of Emesis
Other: Nutritional form inclusion — Food-list form encompassing last 24 hours completion
Other: Blood sampling inclusion — Measurement of biochemical nutrition marker(s); Prealbumin
Other: Intervention at discharge — PUQE-form, nutritional form and Blood sampling
  Groups: Hyperemesis gravidarum

SUMMARY:
This study evaluate the rate of nausea and nutritional status in patients with hyperemesis gravidarum (severe nausea and vomiting in pregnancy) and healthy pregnant women using a questionnaire (PUQE-score), self-reported food/drink intake form and blood test. The Investigators aim for developing normal range of prealbumin measurements (reference values) during first trimester of pregnancy.

DETAILED DESCRIPTION:
Women affected with hyperemesis gravidarum are at severe nutritional risk. Reference values for biochemical parameters evaluating nutritional status during early pregnancy needs to be determined.

The investigators will compare clinical nutritional parameters (weight gain/weight loss) with rate of nausea (PUQE-questionnaire), self-reported nutritional intake form and biochemical measurements (prealbumin) in women admitted to hospital with hyperemesis gravidarum and healthy pregnant women.

For hyperemesis patients measurements will be repeated at discharge.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women < 16 weeks of gestation
* Admitted to hospital for hyperemesis gravidarum (HG group) with nausea and vomiting in pregnancy with at least two of following criteria; weight loss, dehydration, fluid-/electrolyte disturbances, ketonuria

Exclusion Criteria:

* Non-viable pregnancy diagnosed at time of inclusion
* Unable to understand Norwegian
* PUQE-score >= 13 (control group)
* Nausea an vomiting in pregnancy caused by other conditions than Hyperemesis gravidarum

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: * Women admitted to hospital due to Hyperemesis gravidarum
  * Healthy pregnant women (without hyperemesis gravidarum)
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2015-09; Primary Completion 2017-05 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Prealbumin in normal pregnancy | Within 24h at inclusion
  Serum Prealbumin measured during first trimester of pregnancy

SECONDARY OUTCOMES:
Prealbumin related to nutritional parameters | Within 24h at inclusion
  Prealbumin level correlated to PUQE-score and weight change in normal and hyperemesis pregnancies
Change in Prealbumin | Patients will be followed until discharge from hospital, a mean of 5 days, and blood sampling repeated at discharge
  Change in Serum Prealbumin during hospital treatment of hyperemesis gravidarum
Prealbumin in Hyperemesis gravidarum | Within 2h from admission to hospital
  Serum Prealbumin measured when admission to hospital

CONTACTS AND LOCATIONS:
Overall Officials: Jone Trovik, MD, PhD, Principal Investigator — Senior consultant
Locations (1):
- Dpt. of Obstetrics and Gynaecology, Haukeland University Hospital, Bergen, Hordaland, Norway

REFERENCES:
- [Background] Birkeland E, Stokke G, Tangvik RJ, Torkildsen EA, Boateng J, Wollen AL, Albrechtsen S, Flaatten H, Trovik J. Norwegian PUQE (Pregnancy-Unique Quantification of Emesis and nausea) identifies patients with hyperemesis gravidarum and poor nutritional intake: a prospective cohort validation study. PLoS One. 2015 Apr 1;10(4):e0119962. doi: 10.1371/journal.pone.0119962. eCollection 2015. PMID 25830549
- [Background] Stokke G, Gjelsvik BL, Flaatten KT, Birkeland E, Flaatten H, Trovik J. Hyperemesis gravidarum, nutritional treatment by nasogastric tube feeding: a 10-year retrospective cohort study. Acta Obstet Gynecol Scand. 2015 Apr;94(4):359-67. doi: 10.1111/aogs.12578. Epub 2015 Feb 17. PMID 25581215